CLINICAL TRIAL: NCT06282419
Title: The Effect of Visual and Auditory Stimuli Presented to Expectant Fathers on Mothers' Postpartum Breastfeeding Success, Perception of Partner Support and Postpartum Depression
Brief Title: The Effect of Visual and Audio Stimulus Offered to Father-to-be
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Merve Cakil, specialist midwife, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: B.30.2.ATA.0.01.00/542
Record Dates: First submitted 2024-02-02; First posted 2024-02-28 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Ultrasonography Prenatal

STUDY DESIGN:
Intervention Model Description: This is a study that evaluates the effects on mothers by involving fathers in the pregnancy follow-up process through the use of mobile ultrasound.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group 1 (Experimental): Fetal images and fetal heart sound recordings will be taken from the pregnant women in experimental group 1 with a mobile phone compatible portable USG device. Fetal USG images of their babies, taken with a portable USG device, and fetal heart sounds will be sent to the prospective fathers in experimental group 1 by the researcher via WhatsApp application twice a week until birth (at least 3 weeks).
  Interventions: Other: USE OF MOBILE ULTRASOUND
- Experimental group 2 (Placebo Comparator): Fetal USG images and fetal heart sounds taken from the internet, which are not of their babies, will be sent to the prospective fathers by the researcher via WhatsApp application twice a week until birth (at least 3 weeks). In the second stage of the research; Breastfeeding videos prepared by the researcher will be sent to fathers in experimental group 2 twice a week for 4 weeks after birth via WhatsApp application.
  Interventions: Other: ultrasound image taken from the internet
- control group (No Intervention): No visual or auditory stimuli were sent.

INTERVENTIONS:
Other: USE OF MOBILE ULTRASOUND — First stage; Women and their partners who meet the research criteria are at the 32-35th week of pregnancy. was included in the study during the week. First, introductory information forms will be applied to the women and expectant fathers assigned to the experimental and control groups through face-to-face interview technique.
  Then, fetal images and fetal heart sounds will be recorded from the pregnant women in experimental group 1 with a mobile phone compatible portable USG device. Fetal USG images and fetal heart sounds taken with the portable USG device of their babies will be sent to the prospective fathers in experimental group 1 by the researcher via WhatsApp application twice a week until birth (at least 3 weeks). In the second stage of the research; Breastfeeding videos prepared by the researcher will be sent to fathers via WhatsApp twice a week for 4 weeks after birth.
  Arms: Experimental group 1
Other: ultrasound image taken from the internet — First stage; Fetal USG images and fetal heart sounds, not belonging to their babies, taken from the internet, will be sent to the fathers in experimental group 2 via WhatsApp application by the researcher twice a week until birth (at least 3 weeks). In the second stage of the research; Breastfeeding videos prepared by the researcher will be sent to fathers via WhatsApp application twice a week for 4 weeks after birth.
  Arms: Experimental group 2

SUMMARY:
It was aimed to evaluate the effect of visual and auditory stimuli presented to father candidates on postpartum breastfeeding success of mothers, perception of spousal support and postpartum depression. The study, which was carried out in a randomized controlled experimental design, consists of nulliparous pregnant women and their spouses who came to the relevant health center for prenatal control between May 2023 and May 2024. In the study, 132 pregnant women (Experimental group 1:44, Experimental group 2:44, control group:44) were recruited with a priori power analysis. In the study, women and their spouses were assigned to the experimental and control groups by randomization. For randomization, single-group columns between 1-165 were created in the system using the Random Integer Generator method in the Numbers subheading of the random.org website. Considering the numbers 1, 2 and 3 in the column, nulliparous pregnant women coming to the polyclinic were randomly assigned to these numbers. Which numbers constitute which group was determined by drawing lots at the beginning of the research. In data collection, Introductory Information Form for women, Women's Perceived Spousal Support Scale in Early Postpartum Process, Breastfeeding Self-Efficacy Scale-Short Form, Breastfeeding Adaptation Scale and Edinburgh Postpartum Depression Scale; Introductory Information Form for men, Fathers; Breastfeeding Attitude and Participation Scale and Edinburgh Postpartum Depression Scale (for Men) were used. Data; It was evaluated in the SPSS program.

DETAILED DESCRIPTION:
Data were collected by the researcher. The research was conducted in 2 stages. First stage; Women and their partners who meet the research criteria are at the 32-35th week of pregnancy. was included in the study during the week. First, introductory information forms were applied to the women and expectant fathers assigned to the experimental and control groups using the face-to-face interview technique.

Then, fetal images and fetal heart sounds were recorded from the pregnant women in experimental group 1 with a mobile phone compatible portable USG device. Fetal USG images of their babies, taken with a portable USG device, and fetal heart sounds were sent to the expectant fathers in experimental group 1 by the researcher via WhatsApp application twice a week until birth (at least 3 weeks). To the prospective fathers in experimental group 2, fetal USG images and fetal heart sounds taken from the internet, which were not of their babies, were sent by the researcher via WhatsApp application twice a week until birth (at least 3 weeks). At this stage, no intervention was made to the fathers in the control group.

In the second stage of the research; Breastfeeding videos prepared by the researcher were sent to the fathers in experimental groups 1 and 2 via WhatsApp application twice a week for 4 weeks after birth. At this stage, no intervention was made to the fathers in the control group.

At the end of the 4th postpartum week, the women in the experimental groups and the control group were given the Spouse Support Scale Perceived by Women in the Early Postpartum Process, Breastfeeding Self-Efficacy Scale-Short Form, Breastfeeding Adaptation Scale and Edinburgh Postpartum Depression Scale by preparing a Google survey and sending the survey link via WhatsApp application. were provided to fill out.

Likewise, at the end of the 4th postpartum week, the fathers in the experimental groups and the control group were asked to fill out the Fathers; Breastfeeding Attitude and Participation Scale and the Edinburgh Postpartum Depression Scale via a Google survey, and the survey link was sent via WhatsApp application.

Taking USG images: They were taken and recorded by the researcher with a portable USG device. The researcher received a certificate by attending the midwife USG usage course.

Taking fetal heart sounds: They were taken and recorded by the researcher with a portable USG device.

Videos on breastfeeding: Prepared by the research team.

ELIGIBILITY:
Inclusion Criteria:

Criteria for inclusion of pregnant women in the study:

* Being literate
* Being nulliparous
* 32-35. weeks of pregnancy between
* Having a single fetus
* There is no obstacle to vaginal birth
* There is no condition that prevents breastfeeding
* Being open to communication
* Volunteering to participate in the research

Criteria for inclusion of fathers in the study:

* Being literate
* Being over 18 years of age
* Being a father for the first time
* Using a smartphone
* Being open to communication
* Volunteering to participate in the research

Exclusion Criteria:

* Criteria for excluding pregnant women from the study:

  * Illiteracy
  * Having a high risk pregnancy
  * Having a diagnosed psychiatric disease

Exclusion criteria for women in the postpartum period from the study:

* Having given birth prematurely
* Having had a caesarean section
* Development of complications in the mother and/or baby after birth
* A condition that prevents breastfeeding in the mother and/or baby

Criteria for not including fathers in the study:

* Illiteracy
* Being under 18 years of age
* Having a diagnosed psychiatric disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 132 (Estimated)
Dates: Start 2023-08-21 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Introductory Information Form (For Women) | 30 days after birth
  The introductory information form prepared by the researchers consists of 16 questions about the introductory characteristics of women.
Spouse Support Scale Perceived by Women During Early Postpartum Period | 30 days after birth
  The sub-dimensions are named "emotional support" (7 items), "social support" (6 items) and "physical support" (3 items). In the items, 1 was taken as "strongly disagree", 2 as "disagree", 3 as "undecided", 4 as "agree", and 5 as "strongly agree". In negative question items, 1 was taken as "strongly agree", 2 as "agree", 3 as "undecided", 4 as "disagree", and 5 as "strongly disagree".
Breastfeeding Self-Efficacy Scale-Short Form | 30 days after birth
  This scale, which consists of a total of 14 items, is a 5-point Likert type and is evaluated as not at all sure (1 point) and always sure (5 points). The lowest score that can be obtained from the scale is 14 and the highest score is 70. The scale has no cut-off point; a higher score means higher breastfeeding self-efficacy.
Breastfeeding Adaptation Scale | 30 days after birth
  The scale consists of 8 sub-dimensions and 27 items. Scale items are rated on a 5-point Likert scale between 1 point and 5 points (1 point: Strongly disagree, 2 points: Disagree, 3 points: Undecided, 4 points: Agree, 5 points: Strongly agree). Three items in the 6th sub-dimension of the scale, "Discomfort in Breastfeeding", contain negative statements and are rated as 1 (strongly agree) and 5 (strongly disagree). The minimum score that can be obtained from the scale is 27 and the maximum score is 135.
Edinburgh Postpartum Depression Scale | 30 days after birth
  It is a self-evaluation scale consisting of 10 items in four-point Likert format. Responses consisting of four options are scored between 0 and 3, the lowest score that can be obtained from the scale is 0 and the highest score is 30. The cut-off point of EPDS is calculated as 12/13, and women whose total scale score is higher than the cut-off point are considered to be in the risk group.
Introductory Information Form (For Men) | 30 days after birth
  The introductory information form prepared by the researchers consists of 5 questions about the personal characteristics of men.
Fathers' Breastfeeding Attitude and Participation Scale | 30 days after birth
  It consists of a total of 28 items. In this scale, responses are evaluated on a five-point Likert scale: "1 = Strongly disagree", "2 = Disagree", "3 = Undecided", "4 = Agree" and "5 = Strongly agree". The total score to be obtained from the BET subscale varies between 14-70 and the cut-off point of the scale is 58. Those with a total score of ≥58 are considered positive attitudes, and those <58 are considered negative attitudes. The total score to be obtained from the BEK subscale varies between 14-70 and the cut-off point of the scale is 58. Those with a total score of ≥58 are called good participation, and those with <58 are called poor participation.
Edinburgh Postpartum Depression Scale for Men | 30 days after birth
  It is a self-evaluation scale consisting of 10 items in four-point Likert format. Responses consisting of four options are scored between 0 and 3, the lowest score that can be obtained from the scale is 0 and the highest score is 30. The cut-off point of EPDS is calculated as 9/10, and men whose total scale score is higher than the cut-off point are considered to be in the risk group.

CONTACTS AND LOCATIONS:
Overall Officials: Ayla KANBUR, Principal Investigator — Ataturk University
Locations (1):
- Atatürk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No